CLINICAL TRIAL: NCT05575700
Title: Safety of Ibuprofen After Major Orthopaedic Surgeries. The PERISAFE Randomized Clinical Multicentre Trial
Brief Title: Safety of Ibuprofen After Major Orthopaedic Surgeries
Acronym: PERISAFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001CCWL2022
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pain, Acute; Hip Arthropathy; Knee Arthropathy; Safety Issues; Analgesia; Analgesic Adverse Reaction; Postoperative Pain; Postoperative Complications
Keywords: PERISAFE; Hip Arthroplasty; Knee Arthroplasty; Postoperative pain; Analgesia; Safety; Non-steroidal Anti-inflammatory drugs
MeSH Terms: conditions — Acute Pain; Agnosia; Pain, Postoperative; Postoperative Complications | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study medication will be masked by the pharmacy. The experimental medicine will be packed and labelled by Region Hovedstadens Pharmacy in accordance with the Good Manufacturing Practice regulations. The sponsor has a set of sealed, opaque envelopes with the participants' allocation, and these will only be revealed for the investigators when the data has been analysed and abstracts and conclusions covering the different possibilities for interpreting the trial results, have been agreed upon by the steering committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Experimental): Participants received ibuprofen 400 mg tablet administered orally three times daily, with eight hour intervals, for eight days after surgery.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Participants received identical placebo tablet administered orally three times daily, with eight hour intervals, for eight days after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — 400 mg tablet three times daily
  Arms: Ibuprofen
Drug: Placebo — tablet three times daily
  Arms: Placebo

SUMMARY:
Safety of an eight-day treatment with ibuprofen after primary hip and knee arthroplasties.

DETAILED DESCRIPTION:
Hip and knee arthroplasty surgeries are some of the most frequently performed planned procedures in the western world. Multimodal analgesic treatment is the leading analgesic treatment principle, with NSAIDs as an essential part. Ibuprofen, the most frequently prescribed NSAID, is effective in reducing acute postoperative pain. However, ibuprofen may be associated with various serious adverse events, including death, cardiovascular morbidity, gastrointestinal ulcer, and renal impairment. The balance between beneficial and harmful effects of a short-term postoperative treatment with ibuprofen after elective hip and knee arthroplasty is unknown.

Objectives: to assess the adverse events of an eight-day treatment of postoperative pain with ibuprofen in patients undergoing elective primary hip or knee arthroplasty.

Intervention: the participants will be randomized in two groups: a) oral ibuprofen 400 mg 3 times daily for eight days. b) identical oral placebo 3 times daily for eight days.

Design and trial size: PERISAFE is a randomized, placebo-controlled multicentre trial with centralized computer-generated allocation sequence and allocation concealment with unknown block size. Patients, investigators, assessors, caregivers, data-managers, writers of the manuscript, and statisticians will be blinded. A total of 2904 eligible patients are needed to detect or discard an effect corresponding to a relative risk reduction of 1/3 with an acceptable risk of type I error of 5 % and of type II error of 20 %, and a proportion of the composite outcome of serious adverse events of 8% in the experimental group.

Sub-studies:

* Serious adverse events relating to the renal system
* Serious adverse events relating to the cardiovascular system
* Serious adverse events relating to the gastrointestinal system, including major bleeding
* Persistent pain and opioid consumption at 90 days and one year postoperatively. Predictive co-factors include preoperative analgesic treatment, type of anesthesia, gender, age, ASA-classification, diabetes, and type of surgery
* Bayesian re-analysis of the primary and secondary outcomes up to 90 days postoperatively. Further details will appear in the statistical analysis plan
* Health-related quality of life via EQ-5D-5L questionnaire 90-days and one year postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective primary hip and knee arthroplasty.
* Age ≥ 18 years.
* Planned postoperative treatment with NSAID.
* Negative pregnancy test for women in the fertile age.
* Informed consent.

Exclusion Criteria:

* Unable to understand or speak Danish.
* Allergy to or contraindications against ibuprofen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2904 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
A composite outcome of either death, acute myocardial infarction, stroke, pulmonary embolism, deep venous thrombosis, renal failure, major bleeding, re-operation, gastrointestinal ulcer, or readmission within 90 days postoperatively. | Postoperative day 0 to 90.
  Proportion of patients with one or more severe adverse events defined in the composite outcome of either death, acute myocardial infarction, stroke, pulmonary embolism, deep venous thrombosis, renal failure, major bleeding, re-operation, gastrointestinal ulcer, or readmission within 90 days postoperatively.

SECONDARY OUTCOMES:
Hospital free days within 90 days postoperatively. | Postoperative day 0 to 90.
  Days outside the hospital within 90 days postoperatively.
A composite outcome of ibuprofen related adverse events based on an eight-day postoperative diary: dyspepsia, diarrhoea. | Postoperative day 0 to 8.
  Proportion of patients with one or more adverse events of ibuprofen during intervention period, defined as dyspepsia or diarrhoea.
A composite outcome of opioid related adverse events based on an eight-day postoperative diary: nausea, vomiting, constipation, dizziness, confusion, sedation, headache. | Postoperative day 0 to 8.
  Proportion of patients with one or more adverse events of opioid during intervention period, defined as nausea, vomiting, constipation, dizziness, confusion, sedation, or headache.
Health related quality of life questionnaire (EQ-5D-5L) after 90 days | Postoperative day 90.
  Evaluation of health related quality of life via EuroQol five-dimensions 5 point Likert-type scale (EQ-5D-5L) questionnaire, incl. the Euro Visual analogue scales (VAS) from 0-100. 100=the best health you can imagine, 0= the worst health you can imagine.
  The questionnaire of health related quality of life includes: mobility, self-care, usual activities, pain or discomfort, anxiety or depression from a scale of no problems, to slight, moderate, severe problems or unable condition.

OTHER OUTCOMES:
Postoperative pain levels, analgesic treatment, and opioid consumption based on an eight-day postoperative diary. | Postoperative day 0 to 8.
  Pain levels will be measured by Numeric Rating Scale (NRS) from 0-10 (no pain = 0, worst pain = 10). Analgesic treatment including opioid consumption will be indicated in total daily doses in mg.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, Professor, Study Chair — Zealand University Hospital
Locations (11):
- Denmark (11):
  - Private Hospital Gildhøj, Brøndby
  - Bispebjerg Hospital, Copenhagen NV
  - Aalborg University Hospital, Farsø
  - Gentofte Hospital, Hellerup
  - Nordsjællands Hospital Hillerød, Hillerød
  - Zealand University Hospital, Køge
  - Næstved Hospital, Næstved
  - Odense University Hospital, Odense
  - Silkeborg Regional Hospital, Silkeborg
  - Svendborg Hospital, Svendborg
  - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Data will be published anonymised according to ICMJEs (International Committee of Medical Journal Editors) guidelines
Supporting Information: Study Protocol, SAP
Time Frame: Nine month after the trial has ended, and the primary results article has been published
  The study protocol and statistical analysis plan will be available after they have been published. Study protocol will be available at PERISAFE website.
Access Criteria: We will make anonymized data available to other researchers' trough public database such as Zenodo open data repository (CERN), or another equivalent database. Furthermore, researchers wishing to access data from the PERISAFE trial should contact omat@regionsjaelland.dk in the first instance.